CLINICAL TRIAL: NCT02076854
Title: A Novel Motivational Ecological Momentary Intervention for Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F31MH097308 (NIH)
Record Dates: First submitted 2014-02-18; First posted 2014-03-04 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2014-02

CONDITIONS: Eating Disorders
Keywords: eating disorders; anorexia nervosa; treatment; technology
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Text-Message Intervention (Experimental): Participants will undergo four weeks (in a randomized order) of receiving personalized motivational text-messages while receiving CBT for their eating disorder.
  Interventions: Behavioral: Text-Message Intervention
- No Text Message Phase (No Intervention): Participants will receive 4 randomized weeks of not receiving text messages while receiving CBT for their eating disorder.

INTERVENTIONS:
Behavioral: Text-Message Intervention
  Arms: Text-Message Intervention

SUMMARY:
The aim of this study is to pilot an innovative motivational text-message intervention for individuals with anorexia nervosa and subthreshold anorexia nervosa. Patients will receive personalized motivational text-messages as an adjunct to cognitive behavioral therapy (CBT). CBT will be provided to patients at no cost for the duration of the study. The investigators hypothesize that the text-messages will help increase motivation to change and kilocalorie intake and decrease eating disordered behavior.

ELIGIBILITY:
Inclusion Criteria:

* Anorexia nervosa/subthreshold anorexia nervosa (i.e., individuals who exhibit significant dietary restraint)
* 18+ years old

Exclusion Criteria:

* BMI < 16.5
* Medication instability for 6 weeks
* Recent/current suicidal risk
* Comorbid substance abuse or dependence, bipolar disorder, schizophrenia, or mental retardation
* Inability to provide release of information to a medical provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in Motivation to Change Eating Disorder Behaviors | Daily for 8 weeks
Change in Eating Disorder Symptoms | Daily for 8 weeks
Kilocalorie Intake (measured by self-report food records) | Daily for 8 weeks

SECONDARY OUTCOMES:
Feasibility measured by compliance with daily questionnaire | 8 weeks
Acceptability measured by self-report ratings | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Eating Disorders Program, Boston University, Boston, Massachusetts, United States